CLINICAL TRIAL: NCT03461042
Title: The Placebo Controlled Randomized Double Blind Multicenter Study to Investigate Effectiveness and Safety of Combination Use of Melatonin Receptor Agonist for Dose Reduction or Interruptions of BZD and Non-BZD Hypnotics on Chronic Insomnia
Brief Title: The Study of Combination Use of Melatonin Receptor Agonist for Dose Reduction or Interruptions of Benzodiazepine (BZD) and Non-BZD Hypnotics on Chronic Insomnia
Acronym: BRED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Yoyogi Sleep Disorder Clinic, Foundation of Sleep and Health Science (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 293/CR1-003 / TRIPSYCHI1407
Record Dates: First submitted 2018-02-14; First posted 2018-03-09 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2021-01

CONDITIONS: Chronic Insomnia
Keywords: Chronic insomnia; Ramelteon; Rozerem; dose reduction
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm R (Experimental): Co-administer following medication for 12 weeks since informed consent; R group: taking capsule of Ramelteon 8mg once daily before sleeping.
  Interventions: Drug: Ramelteon 8mg
- Arm PL (Placebo Comparator): Co-administer following medication for 12 weeks since informed consent; Placebo group: taking capsule of Placebo once daily before bedtime.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon 8mg — Ramelteon 8mg once daily before bedtime for 12 weeks since informed consent
  Arms: Arm R
Drug: Placebo — Placebo capsule once daily before bedtime for 12 weeks since informed consent
  Arms: Arm PL

SUMMARY:
To investigate effects on combination use of Ramelteon in the dose reduction or interruption process of (non-)BZD hypnotics during the dose reduction or interruption algorithm.

DETAILED DESCRIPTION:
The hypnotic 'Ramelteon' does not have effect on Gamma Aminobutyric Acid (GABA-A) receptor that relates to the formation of addiction to the BZD or non-BZD hypnotics. Some results of clinical trials has been reported that the dose reduction or interruption of (non-)BZD hypnotics was achieved on combination use of Ramelteon by using its characteristic of the action mechanism with safely and effectively. However, these results have not been confirmed with randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting Criteria 1 or 2 and Criteria 3 and all subsequent criteria will be included in the study:

1. Patients diagnosed as chronic insomnia having sleep onset disturbance, and with a duration of the disease of at least 6 months
2. Patients diagnosed with chronic insomnia comorbid with mood disorders (depression or bipolar disorder) can be included to this study if they have remission of mood symptoms.
3. Patients taking (non-)BZD hypnotics (including etizolam at bedtime) at a fixed dose in the following patterns since at least 1 month prior to consent (over 90% of drug compliance should be confirmed at the time of medical interview):

   * Patients taking 2 drugs at the usual dose (1 unit)
   * Patients taking 3 drugs at the usual dose (1 unit)
   * Patients taking 4 drugs at the usual dose (1 unit)
   * Patients taking a drug at 2-fold of the usual dose (2 units)
   * Patients taking a drug at 2-fold of the usual dose (2 units) and a drug at the usual dose (1 unit)
   * Patients taking a drug at 2-fold of the usual dose (2 units) and 2 drugs at the usual dose (1 unit)
   * Patients taking 2 drugs at 2-fold of the usual dose (2 units) Patients whose total dosage are 2～4 units of 1～4 drugs can be also included. But attention needed not to conflict with exclusion criteria 2.

     ※Dosage cannot exceeded 2 units per 1 drug.
   * Patients whose symptoms of insomnia were stabilized, and the investigators determined that the (non-) BZD hypnotics could be reduced or discontinued
   * Patients aged 20 years or older at the time of consent
   * Patients who are willing to comply with algorithm for dose reduction and discontinuation
   * Patients who can understand the content of the study and provide consent to participate in the study in writing on their own will.

Exclusion Criteria:

Subjects meeting any of the following criteria will not be included in the study:

* Patients with secondary insomnia
* Patients taking (non-)BZD hypnotics at a dose exceeding 2-fold of the usual dose
* Patients taking barbiturate and non-barbiturate hypnotics and Suvorexant.
* Patients taking hypnotics other than medicinal pharmaceuticals (including Over The Counter (OTC), supplements believed to be effective for insomnia and melatonin )
* Patients taking mianserin hydrochloride, mirtazapine, and trazodone hydrochloride
* Patients taking antipsychotics
* Patients taking anxiolytic or clonazepam at bedtime

  *Patient taking anxiolytic and/or clonazepam at times except for bed-time will be included in the study. However, dosage and timing of administration can not be changed during the study period.
* Patients who took ramelteon within 1 month prior to the informed consent
* Patients in whom the dose of psychotropics except for the items 2～7 were changed within 1 month prior to the informed consent
* Patients who are comorbid with depression or bipolar disordered and in whom depressive symptoms have not remitted
* Patients in whom frequency in Q9 of PHQ "thoughts that you would be better off dead or thoughts of hurting yourself in some way" is "more than half the days (in the past 2 weeks)" or the total score is 10 or higher
* Patients with dementia, schizophrenia, drug dependence and alcoholic
* Patients with liver/kidney disorder, female subjects who are pregnant or in breast-feeding, and malignant neoplasm
* Night workers
* Patients meeting contraindications for ramelteon
* Other patients judged ineligible for participation in the study by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
The achievement ratio of the 50% dose reduction of (non-)BZD hypnotics (Diazepam conversion value) at 12weeks or withdrawal without any deterioration of insomnia symptoms. | 12 weeks
  Evaluate the achievement ratio of the 50% or more of dose reduction by Participant's diary
The rate of subjects who achieved more than 50% dose reduction of (non-)BZD hypnotics (Diazepam conversion value) at 12 weeks or withdrawal since informed consent. | 12 weeks
  The rate of subjects who achieved more than 50% of dose reduction (Diazepam conversion value) will be assessed by Participant's diary

SECONDARY OUTCOMES:
The achievement ratio of the 50% dose reduction (Diazepam conversion value) at 4weeks and 8weeks | at 4 weeks and 8weeks
  The rate of subjects who achieved more than 50% dose reduction (Diazepam conversion value) will be assessed by Participant's diary
The average of the dose reduction rate at 4weeks, 8weeks and 12weeks | at 4 weeks, 8weeks and 12 weeks
  The average of the dose reduction rate will be assessed by Participant's diary
The achievement ratio of the 100% dose reduction at 12weeks or withdrawal | 12 weeks
  The achievement ratio of the 100% dose reduction will be assessed by Participant's diary
The variation in total score of Pittsburg Sleep Quality Index (PSQI) at 4weeks, 8weeks and 12weeks | at 0, 4, 8 and 12 weeks
  The variation in total score of PSQI will be assessed by the PSQI value sets sets at week 0, 4, 8 and 12. (The range of total score is 0-21. Higher scores represent worse tendency of the symptoms.)
The variation in total score of Athens Insomnia Scale (AIS) at 4weeks, 8weeks and 12weeks | at 0, 4, 8 and 12 weeks
  The variation in total score of AIS will be assessed by the AIS value sets at week 0, 4, 8 and 12. (The range of total score is 0-24. Higher scores represent worse tendency of the symptoms.)
The variation in Patient health questionnaire (PHQ-9) score at 4weeks, 8weeks and 12weeks | at 0, 4, 8 and 12 weeks
  The variation in PHQ-9 score will be assessed by the PHQ-9 value sets at week 0, 4, 8 and 12. (The range of total score is 0-27. Higher scores represent worse tendency of the symptoms.)
Guide to the use of the clinical withdrawal assessment scale for benzodiazepines (CIWA-B) score at 4weeks, 8weeks and 12weeks | at 4, 8 and 12 weeks
  The variation in CIWA-B (Guide to the use of the clinical withdrawal assessment scale for benzodiazepines) score will be assessed by the CIWA-B value sets at week 4, 8 and 12. (The range of total score is 0-80. Higher scores represent worse tendency of the symptoms.)
Patient global impression of therapy (PGI) score at 12weeks or withdrawal | 12 weeks
  PGI(Patient global impression of therapy) score will be assessed by the PGI value sets at 12weeks or withdrawal. (The range of total score is 0-21. Higher scores represent worse tendency of the symptoms.)
The variation in Ben-dep(Benzodiazepine Dependence Self-Report Questionnaire) score at 12weeks or withdrawal | at 0 and 12 weeks
  The variation in Ben-dep score will be assessed by the Ben-dep value sets at 0 and 12weeks or withdrawal. (The range of total score is 0-100. Higher scores represent worse tendency of the symptoms.)
Adverse Events | 12 weeks
  Adverse Events will be determined by the latest version of MedDRA/J （Medical Dictionary for Regulatory Activities/J).

CONTACTS AND LOCATIONS:
Overall Officials: Yuichi Inoue, MD, Ph.D., Principal Investigator — Yoyoghi Sleep Disorder Clinic / Foundation of Sleep and Health Science
Locations (1):
- Yoyogi Sleep Disorder Clinic, Foundation of Sleep and Health Science, Shibuya-ku, Tokyo, Japan